CLINICAL TRIAL: NCT04311190
Title: Family ENgagement in Intensive Care Environments (FENICE): a Quasi-experimental Study
Brief Title: Family Engagement in Intensive Care Unit
Acronym: FENICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Udine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3070
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Critical Care; Intensive Care Unit; Nurse's Role; Family Members

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICU A (Experimental): Family members' involvement in the care of their beloved one
  Interventions: Other: Family engagement
- ICU B (No Intervention): Standard care

INTERVENTIONS:
Other: Family engagement — Physical exercises and simple care tasks
  Arms: ICU A

SUMMARY:
We hypothesized that engaging families in the care of critically ill patients could improve outcome both at the family and at the patient levels. Thus, the aim of this project is to assess the effects of a family engagement program on family members' satisfaction and on patients' well-being and quality of life.

DETAILED DESCRIPTION:
Despite the health care professionals should consider the active involvement of families in Intensive Care Unit (ICU), little research investigating family member's contributions to care, including its outcomes on family itself and on patient care, has been rendered available. To assess the effects of a family engagement program on family members' satisfaction and on patients' well-being and quality of life. A quasi-experimental study with two non-randomized groups (94 per each group) will be performed in two general ICUs of an Academic Italian Hospital. The intervention will be carried out in a single ICU and consists of family members' involvement in the care of their beloved one with bed physical exercises and simple care tasks. Participants will be assessed for outcomes including the family satisfaction, assessed with the FS-ICU tool within 48 hours after the patient's discharge from ICU, the patient's sense of well-being, measured with a visual analogue scale within 30 minutes after the time period of a visit, and the quality of life, investigated with the SF-12 questionnaire within the first 48 hours after admission in ICU, at three and six months after ICU discharge by telephone. First, this study constitutes a significant step in a research agenda aimed at deepening the nursing sensitive outcomes in ICUs and the quality of hospital care. Secondly, result from this study may have the potential to better understand how families may modify patients' outcomes and whether the family members would benefit from an engagement program.

ELIGIBILITY:
Inclusion Criteria:

PATIENT

* 18 years of age and older;
* expected to stay in-ICU at least three days;
* with high or low acuity conditions.

FAMILY MEMBER

* being the patient's spouse, or in a blood relation, or next of kin, and/or with whom the patient spends most of the time;
* 18 of age or above;
* willing to visit the patient on a daily basis;
* willing to participate in the study.

Exclusion Criteria:

PATIENT Patients' discharge from ICU, transfer to another hospital, or death.

FAMILY MEMBER The unexpected suspension of visiting their loved ones in ICU daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Family satisfaction (FS) | Within 48 hours after the patient's discharge from ICU
  FS-ICU tool

SECONDARY OUTCOMES:
Patient's sense of well-being | 30 minutes after the family involvement for the intervention group and in the same hours after the ICU visiting hours for the control group
  Visual analogue scale
Quality of Life (QoL) | At three and six months after ICU discharge
  SF-12

CONTACTS AND LOCATIONS:
Overall Officials: Amato De Monte, Study Chair — Department of Anestesia and Intensive Care (ASUFC) - UDINE, IT

IPD SHARING:
Plan to Share IPD: No